CLINICAL TRIAL: NCT03125174
Title: Characterization of Airway Mucus in Bronchiectasis Patients and Healthy Controls
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: 16-3142
Record Dates: First submitted 2017-04-14; First posted 2017-04-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Bronchiectasis Adult
Keywords: sputum; bronchiectasis; lung disease
MeSH Terms: conditions — Bronchiectasis; Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — sputum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control: healthy individuals with no history of lung disease
- bronchiectasis patients: individuals with a diagnoses of bronchiectasis

SUMMARY:
Analysis of mucus, mucin and DNA concentration, MUC5B/5AC ratio, rheology, osmotic pressure, cohesion and nucleotides in sputum on 30 individual samples of good quality in healthy individuals and those with bronchiectasis. (60 total)

DETAILED DESCRIPTION:
In this study the investigators will investigate the mucus properties in individuals with idiopathic bronchiectasis and healthy individuals without a history of lung disease. In order to understand how mucus is abnormal in disease conditions, the investigators need to understand the mucus biochemical and biophysical properties in healthy individuals. In this study the investigators will prospectively recruit patients with bronchiectasis and healthy individuals from the community to provide airway sputum samples. In these samples the investigators will measure an array of mucus properties. This will help our understanding of the mucus-obstructive lung diseases and facilitate the development of appropriate and effective disease prevention strategies.

A key question is whether mucus is hyper-concentrated and has abnormal biophysical properties in individuals with mucus-obstructive lung disease. To answer this question, the investigators need to understand the properties of the mucus in individuals with idiopathic bronchiectasis and no history of lung disease. This study will allow us to collect airway mucus (sputum) from individuals with bronchiectasis and healthy individuals with no history of lung disease.

ELIGIBILITY:
Participants who meet all the following criteria are eligible for the study:

* Written informed consent
* Bronchiectasis patients: Available CT of the chest that shows evidence of dilated airways fulfilling radiographic criteria for bronchiectasis in more than one lobe and chronic cough.

Participants who meet any of the following criteria will not be eligible for the study:

* Healthy individuals: A history of lung disease, current asthma symptoms or medication use, premature birth (<37 week gestation), a history of lung disease of infancy, or neurological or cardiovascular illness, current smoker or a history of smoking tobacco products.
* Bronchiectasis patients: Premature birth (<37 week gestation), a history of lung disease of infancy, or neurological or cardiovascular illness.
* Younger than 18 years of age

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The proposed study will recruit 30 patients with bronchiectasis and 30 healthy individuals with no history of lung disease aged over the age of 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2017-06-27 (Actual); Study Completion 2017-06-27 (Actual)

PRIMARY OUTCOMES:
Mucus concentration (% solids) | 6 months
  The percentage of solid content of sputum (an index of hydration) will be calculated my measuring the wet to dry weight ratio using a microbalance (mean percent solids ± standard deviation).

SECONDARY OUTCOMES:
Biophysical properties of mucus by rheology | 6 months
  The rheological properties of the sputum will be assayed by macro-rheology (cone and plate) and microbead rheology. Macro-rheology provides measures of the viscosity (median log viscosity in Pascal (range)) and elasticity (median log elasticity in Pascal (range) of the sputum. Microbead rheology is performed by analyzing the diffusive motion of embedded 1μm tracer particles (6). The primary outcome measure from microbead rheology will be the mean square displacement MSD(Mean squared displacement) (median MSD cm2 s-1 (range)).
Mucin composition by mass spectroscopy | 6 months
  We will use mass spectroscopy to determine the relative abundance of the two major polymeric mucin proteins, MUC5B(Mucin type 5B)and MUC5AC(Mucin type 5AC), which are responsible for the viscoelastic properties of mucus.
Sputum extracellular nucleotide analysis | 6 months
  Sputum adenosine and adenine nucleotides will be ethenoderivatized and measured by HPLC(High performance liquid chromatography) analysis (7) (median nucleotide concentration in μg/ml (range)).
Osmotic Pressure | 6 months
  The osmotic pressure of the mucus will be assessed by placing an aliquot of mucus onto an osmometer with a 10kDa (10 kilodaltons) molecular weight polyethersulfone membrane (Millipore) separating the test chamber and reference chamber filled with PBS (phosphate-buffered saline) (mean osmotic pressure in Pascal ± standard deviation).
Total mucin concentration | 6 months
  Mucins will be quantitated using sepharose CL2B(Cross-linked derivative of Sepharose 2B) UPLC(Ultra performance liquid chromatography) coupled to an Optilab interference refractometer with a filter at 680 nm and parallel flow chambers for solvent and the solution (mean mucin concentration (μg/ml) ± standard deviation) (4). With this approach, we will ensure that the solute is at full Donnan equilibrium with the solution within the context of gel chromatography, which creates an accurate equilibration of solute and solvent. This procedure also separates the mucins from contaminating proteins, allowing the mucins to be isolated for biochemical studies. DNAse can be added if significant DNA is present.
polymeric DNA concentration | 6 months
  The quantification of free DNA will be performed using the DNA Quant-iT PicoGreen assay (Molecular Probes, Inc., Eugene, OR, USA), which utilizes an ultra-sensitive fluorescent nucleic acid stain for quantitating double-stranded DNA (median log DNA concentration (μg/ml) (range)).

CONTACTS AND LOCATIONS:
Overall Officials: Richard Boucher, MD, Study Chair — University of North Carolina, Chapel Hill; Kathryn Ramsey, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - Center for Environmental Medicine Asthma and Lung Biology, Chapel Hill, North Carolina
  - Marsico Research Institure at Meadowmont, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No